CLINICAL TRIAL: NCT02534636
Title: Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986165 in Healthy Subjects and to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Efficacy of BMS-986165 in Subjects With Moderate to Severe Psoriasis
Brief Title: Safety Study of BMS-986165 in Healthy Subjects and to Treat Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: IM011-002
Record Dates: First submitted 2015-08-23; First posted 2015-08-27 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — deucravacitinib; Interferon alpha-2; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: Single ascending dose (Experimental): BMS-986165 or Placebo specified dose on specified days
  Interventions: Drug: BMS-986165; Other: Placebo
- Part B: Multiple ascending dose (Experimental): BMS-986165 or Placebo + Interferon alpha-2a recombinant specified dose on specified days
  Interventions: Drug: BMS-986165; Drug: Interferon alpha-2a recombinant; Other: Placebo
- Part C: Multiple ascending dose (Experimental): BMS-986165 or Placebo specified dose on specified days
  Interventions: Drug: BMS-986165; Other: Placebo
- Part D: Relative Bioavailability (Experimental): BMS-986165 (Liquid) + BMS-986165 (Capsule) + Famotidine specified dose on specified days
  Interventions: Drug: BMS-986165; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986165
Drug: Interferon alpha-2a recombinant
  Arms: Part B: Multiple ascending dose
Drug: Famotidine
  Arms: Part D: Relative Bioavailability
Other: Placebo
  Arms: Part A: Single ascending dose; Part B: Multiple ascending dose; Part C: Multiple ascending dose

SUMMARY:
The purpose of this study is to establish if BMS-986165 is safe and effective at treating autoimmune diseases. BMS-986165 which has shown some promise in preclinical studies for inhibiting autoimmune conditions. This study will be the first time this drug is given to humans, and will be conducted entirely in healthy subjects. It will be run in 4 Parts. Part A will investigate single oral doses of drug. Part B will investigate giving the drug daily for 14 days. Part C will investigate daily doses for 14 days in healthy volunteers with Japanese decent. Part D will investigate whether food, stomach acidity or giving the drug in a capsule makes a difference to the safety and potential use of this drug.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy Male and Female participants
* 18 to 50 years of age (Parts A-D)

Exclusion Criteria:

* Participants that had recent infections
* Participants with low blood pressure or increased heart rate
* Participants with any chronic health related problems
* Participants with active cancer within the last 5 years
* Participants with any other major medical illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety of a single oral dose of BMS-986165 based on number of incidence of AE, SAEs, AEs leading to discontinuation or death, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Approximately 3 months
  Adverse Event (AE), Serious adverse event (SAE)
Tolerability of a single oral dose of BMS-986165 based on number of incidence of AE, SAEs, AEs leading to discontinuation or death, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Approximately 3 months
Safety of a multiple oral dose of BMS-986165 based on number of incidence of AE, SAEs, AEs leading to discontinuation or death, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Approximately 3 months
Tolerability of a multiple oral dose of BMS-986165 based on number of incidence of AE, SAEs, AEs leading to discontinuation or death, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Approximately 3 months

SECONDARY OUTCOMES:
Effect of BMS-986165 on electrocardiographic (ECG) parameters such as heart rate in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months
Effect of BMS-986165 on electrocardiographic (ECG) parameters such as PR interval in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months
Effect of BMS-986165 on electrocardiographic (ECG) parameters such as QRS interval in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months
Effect of BMS-986165 on electrocardiographic (ECG) parameters such as QTc interval in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Catlett IM, Aras U, Hansen L, Liu Y, Bei D, Girgis IG, Murthy B. First-in-human study of deucravacitinib: A selective, potent, allosteric small-molecule inhibitor of tyrosine kinase 2. Clin Transl Sci. 2023 Jan;16(1):151-164. doi: 10.1111/cts.13435. Epub 2022 Nov 22. PMID 36325947
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx